CLINICAL TRIAL: NCT00315159
Title: Conservative Management With Isolated Sentinel Lymph Node Biopsy in Vulvar Cancer Patients With Sentinel Lymph Nodes Determined to be Negative for Metastatic Disease.
Brief Title: Conservative Management With Isolated Sentinel Lymph Node Biopsy in Vulvar Cancer Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Richard G. Moore, MD, Richard Moore, M.D., Women and Infants Hospital of Rhode Island
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-0031
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Vulvar Cancer
Keywords: Squamous; Cell; Carcinoma; Vulva; Sentinel Node
MeSH Terms: conditions — Vulvar Neoplasms; Carcinoma | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- No intervention (No Intervention): Patients with negative SLN will be followed on no intervention arm
  Interventions: Procedure: Sentinel Node Biopsy

INTERVENTIONS:
Procedure: Sentinel Node Biopsy — Inguinal sentinel node biopsy will be performed.

SUMMARY:
The purpose of this study is to evaluate a less invasive procedure for the evaluation of the inguinal (groin) nodes in patients with a primary squamous cell carcinoma of the vulva. Each patient will undergo a sentinel lymph node dissection as well as resection of the primary tumor on the vulva. Patients who are determined to have sentinel nodes that are negative for metastatic disease will not receive a full groin dissection. Patients who have sentinel lymph nodes that contain metastasis will undergo a complete inguinal dissection. The study will evaluate the long-term outcomes in patients who receive only a sentinel lymph node dissection without a complete dissection. All patients entered onto the study will have a biopsy proven squamous cell carcinoma of the vulva. Each patient will be enrolled by a Gynecologic Oncologist practicing out of Women & Infants Hospital

DETAILED DESCRIPTION:
Conservative Management with Isolated Sentinel Lymph Node Biopsy in Vulvar Cancer Patients with Sentinel Lymph Nodes Determined to be Negative for Metastatic Disease.

Introduction The American Cancer Society estimates there will be 4000 new cases of vulvar cancer for the year 2003(1). The majority of these patients will undergo surgical therapy with groin node dissection to assess the inguinal nodal chain for evidence of metastatic disease. For many years there has been a search for a less radical surgical approach to evaluating the inguinal lymphatic basin. The classic approach to vulvar cancer was an en-bloc resection of the vulva and groins with a single incision. This approach led to complication rates as high as 69% for chronic leg edema and 85 % for wound breakdown(2). In an effort to reduce the morbidity of groin node dissections, the triple incision technique was introduced(3). A GOG study evaluating limited surgery with wide local excision and superficial groin node dissection reported rates of chronic lymphedema of 19% and wound infection and or separation of 29%(4). In their report on penile carcinoma the concept of a sentinel node as the first group of nodes in the inguinal lymphatic chain was put forth by Cabanas et al.(5). Morton and colleagues advanced the technique of sentinel node lymphatic mapping in patients with cutaneous melanoma(6). In 1994 Levenback et al, described of the use of isosulfan blue dye for the detection of sentinel nodes in the inguinal lymphatic chain(7). To date, a number of studies have been performed evaluating the utility of sentinel node technology and its application in vulvar malignancies (Table 1)(7-20). For melanoma, the sentinel node dissection has become the standard of care for the evaluation of the lymphatic basins. Many cancer centers, including Women and Infants' Hospital, use sentinel node dissection for the evaluation of axillary nodes in breast cancer patients as their standard of care. This technology has decreased the rate of chronic arm edema in breast cancer patients.

Inguinal node metastasis in patients with squamous cell carcinoma of the vulva is reported to be as high as 27%(21). Consequently, a large number of patients may undergo a potentially morbid procedure without any gain. Non-invasive methods for the evaluation of the inguinofemoral nodes such as CT, MRI and PET scans have not yet been proven reliable. Sentinel node biopsy utilizing Tc-99m sulfur colloid and isosulfan blue dye allows for evaluation of nodal status in patients with vulvar malignancies through minimally invasive surgery. Our study, at Women and Infants' Hospital, employed Tc-99m sulfur colloid and isosulfan blue dye to identify sentinel nodes in the inguinal lymphatic chain of patients with primary squamous cell carcinoma of the vulva. Twenty nine patients were enrolled and 107 sentinel nodes were studied with no false negative SLN being reported(22) There are over 175 patients in the reported literature who have undergone a SLN dissection for the evaluation of the inguinal lymphatic basin for metastatic disease. To date there have been no false negative SLN reported. We feel the SLN dissection has been proven to be reliable and safe procedure both at our institution and others around the world. Further studies need to be performed in order to evaluate the use of SLN dissection alone in patients with pathologic negative sentinel nodes for metastasis. This study will evaluate the use of sentinel node dissection alone and management of these patients who potentially do not need or will benefit from a full inguinal node dissection.

Sentinel Node Concept Sentinel node dissection was first applied for the evaluation of inguinal nodal basins in patients with penile cancer(23). The sentinel node concept is based on the belief that certain anatomical areas are drained by individual nodal chains with the first lymph node in this chain being the sentinel node. It has been shown the sentinel node is predictive of the status of the lymphatic basin for the presence of metastatic disease to non-sentinel nodes. The use of both lymphazurin blue dye and technetium-99m sulfur colloid has been shown to reliably identify sentinel nodes in many cancers such ad melanoma, breast and colon. This technology has also been studied in patients with vulvar malignancies and has been shown to detect a sentinel node 100% of the time(22). With a limited number of sentinel nodes obtained from a lymphatic basin a more complete pathologic evaluation of the lymph node can be performed. The use of ultra-staging (serial sectioning) allows for smaller metastasis and micrometastasis to be reliably detected. Sentinel lymph node technology will allow for a more complete surgical and pathologic evaluation of the inguinal lymphatic basins with a potential benefit of avoiding a complete inguinal node dissection for patients with a SLN determined to be negative for metastatic disease.

Study Design

This is a prospective trial examining conservative management of patients with inguinal sentinel nodes that have been deemed negative for metastatic disease in patients with primary squamous cell carcinoma of the vulva.

Number of Patients:

The goal of this study is to enroll 100 patients over a 5 year period and follow each for a total of three years.

Sentinel Lymph Node Technique:

Each patient will undergo two intradermal peritumoral injections with a total of 2-3 mCi of unfiltered technetium-99m sulfur colloid in a volume of 1cc, within 24 hours prior to surgery. These injections will take place in the nuclear medicine suite at Rhode Island Hospital under Dr. Richard Noto's supervision. Following the injection of the Tc-99m sulfur colloid a lymphoscintigram will be performed to detect the presence of a sentinel node. Intra-operatively, 5 to 10 minutes prior to the groin dissection, 3 cc of isosulfan blue dye will be injected at the peritumoral edge in a manner and location similar to the Tc-99m sulfur colloid injection. An inguinal dissection will then performed before the radical excision of the vulvar tumor. Prior to the groin node incision, a hand held collimated gamma counter will be used to identify the location of the sentinel node. This area will be marked with ink on the skin surface. An inguinal incision will be made and the inguinal lymphatic beds will be dissected to identify blue afferent lymphatic tracts and/or blue stained lymph nodes. A hand held collimated gamma counter will be used to detect any lymph nodes with increased activity, defined as a count greater than 5 % of that at the injection site, through the groin incision. Also, any lymph node with a blue lymphatic tract leading to it or stained blue will be considered a sentinel node. As well, any lymph node identified with the hand held gamma counter as taking up the Tc-99m sulfur colloid will be considered a hot sentinel node. Each sentinel node will be evaluated with a 10 second gamma count and labeled as hot and blue, hot and non-blue or cold and blue. With completion of the sentinel node groin node dissection, the lymphatic beds will be re-scanned with the gamma counter to ensure all sentinel nodes have been removed. Once the SLN groin dissection is complete the incision will be closed and a full groin dissection will be done at a separate sitting pending the pathologic evaluation of the sentinel lymph node. The remainder of the surgery for the treatment of the primary tumor will then be completed with a current standard of care procedure depending on the size and location of the tumor.

Pathologic Analysis of Sentinel Lymph Nodes:

Each sentinel lymph node will be serially sectioned at 2mm intervals parallel to the long axis and totally submitted for histologic evaluation in one or more blocks. From each block, five slides will be cut at 100 micron intervals and stained with hematoxylin and eosin. A parallel slide at each level will be cut and held for batch cytokeratin AE1/AE3 immunohistochemical staining if negative for metastasis by initial H&E staining. The largest dimension of each metastasis will be measured and recorded in order to track the presence of micrometastasis defined as a metastatic focus less than 2mm in size.

Patient Management Protocol:

Patients enrolled on to the sentinel lymph node protocol will undergo a sentinel lymph node dissection as described above followed by a radical excision of the primary tumor. Patients with sentinel nodes found to contain metastatic disease from the primary vulvar malignancy will under go a complete inguinal lymph node dissection as per standard care. Patients with sentinel lymph nodes deemed negative for metastatic disease based on ultra-staging and H&E staining will be followed with conservative management (no further groin node dissection). Each of these patients will be followed clinically at 3 month intervals for the first three years for a total study follow up period of three years. Any patient determined to have a groin recurrence will be treated with current standard of care modalities as appropriate for their recurrence. Published data documenting a 5-7% unanticipated groin failures in patients with negative lymphadenectomies will be used as the comparative outcomes (25).

ELIGIBILITY:
Inclusion Criteria:

1. Patient of any age 18 years or over.
2. Biopsy proven squamous cell carcinoma of the vulva.
3. Depth of invasion 1mm or greater.
4. Patients with groins clinically negative for nodal metastasis.
5. Patients that are candidates for groin dissections.

Exclusion Criteria:

1. Any patient below the age of 18
2. Patients with clinically suspicious groin nodes for metastatic disease.
3. Patients with non-squamous cell vulvar lesions.
4. Depth of invasion less than 1mm.
5. Patients refusing to sign an informed consent form.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2003-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Determination of inguinal recurrence rates in patients with negative sentinel lymph node biopsy alone. | Three years

SECONDARY OUTCOMES:
Ability to detect inguinal sentinel nodes in vulvar cancer patients. | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Richard G Moore, MD, Principal Investigator — Women and Infants' Hospital
Locations (1):
- Women and Infants' Hospital of Rhode Island, Providence, Rhode Island, United States

REFERENCES:
- [Background] Jemal A, Murray T, Samuels A, Ghafoor A, Ward E, Thun MJ. Cancer statistics, 2003. CA Cancer J Clin. 2003 Jan-Feb;53(1):5-26. doi: 10.3322/canjclin.53.1.5. PMID 12568441
- [Background] Jemal A, Murray T, Ward E, Samuels A, Tiwari RC, Ghafoor A, Feuer EJ, Thun MJ. Cancer statistics, 2005. CA Cancer J Clin. 2005 Jan-Feb;55(1):10-30. doi: 10.3322/canjclin.55.1.10. PMID 15661684
- [Background] Podratz KC, Symmonds RE, Taylor WF, Williams TJ. Carcinoma of the vulva: analysis of treatment and survival. Obstet Gynecol. 1983 Jan;61(1):63-74. PMID 6823350
- [Background] Hacker NF, Leuchter RS, Berek JS, Castaldo TW, Lagasse LD. Radical vulvectomy and bilateral inguinal lymphadenectomy through separate groin incisions. Obstet Gynecol. 1981 Nov;58(5):574-9. PMID 7301232
- [Background] Cabanas RM. An approach for the treatment of penile carcinoma. Cancer. 1977 Feb;39(2):456-66. doi: 10.1002/1097-0142(197702)39:23.0.co;2-i. PMID 837331
- [Background] Morton DL, Wen DR, Wong JH, Economou JS, Cagle LA, Storm FK, Foshag LJ, Cochran AJ. Technical details of intraoperative lymphatic mapping for early stage melanoma. Arch Surg. 1992 Apr;127(4):392-9. doi: 10.1001/archsurg.1992.01420040034005. PMID 1558490
- [Background] Levenback C, Burke TW, Morris M, Malpica A, Lucas KR, Gershenson DM. Potential applications of intraoperative lymphatic mapping in vulvar cancer. Gynecol Oncol. 1995 Nov;59(2):216-20. doi: 10.1006/gyno.1995.0011. PMID 7590476
- [Background] Levenback C, Morris M, Burke TW, Gershenson DM, Wolf JK, Wharton JT. Groin dissection practices among gynecologic oncologists treating early vulvar cancer. Gynecol Oncol. 1996 Jul;62(1):73-7. doi: 10.1006/gyno.1996.0192. PMID 8690296
- [Background] Levenback C. Intraoperative lymphatic mapping and sentinel node identification: gynecologic applications. Recent Results Cancer Res. 2000;157:150-8. doi: 10.1007/978-3-642-57151-0_13. PMID 10857169
- [Background] Levenback C, Coleman RL, Ansink A, van der Zee AG. Re: Terada et al.: Sentinel node dissection and ultrastaging in squamous cell cancer of the vulva. Gynecol Oncol 76:40-44, 2000. Gynecol Oncol. 2000 Jun;77(3):484-5. doi: 10.1006/gyno.2000.5832. No abstract available. PMID 10831370
- [Background] Levenback C, Coleman RL, Burke TW, Bodurka-Bevers D, Wolf JK, Gershenson DM. Intraoperative lymphatic mapping and sentinel node identification with blue dye in patients with vulvar cancer. Gynecol Oncol. 2001 Nov;83(2):276-81. doi: 10.1006/gyno.2001.6374. PMID 11606084
- [Background] Decesare SL, Fiorica JV, Roberts WS, Reintgen D, Arango H, Hoffman MS, Puleo C, Cavanagh D. A pilot study utilizing intraoperative lymphoscintigraphy for identification of the sentinel lymph nodes in vulvar cancer. Gynecol Oncol. 1997 Sep;66(3):425-8. doi: 10.1006/gyno.1997.4798. PMID 9299256
- [Background] Terada KY, Coel MN, Ko P, Wong JH. Combined use of intraoperative lymphatic mapping and lymphoscintigraphy in the management of squamous cell cancer of the vulva. Gynecol Oncol. 1998 Jul;70(1):65-9. doi: 10.1006/gyno.1998.5035. PMID 9698476
- [Background] de Hullu JA, Doting E, Piers DA, Hollema H, Aalders JG, Koops HS, Boonstra H, van der Zee AG. Sentinel lymph node identification with technetium-99m-labeled nanocolloid in squamous cell cancer of the vulva. J Nucl Med. 1998 Aug;39(8):1381-5. PMID 9708512
- [Background] Echt ML, Finan MA, Hoffman MS, Kline RC, Roberts WS, Fiorica JV. Detection of sentinel lymph nodes with lymphazurin in cervical, uterine, and vulvar malignancies. South Med J. 1999 Feb;92(2):204-8. doi: 10.1097/00007611-199902000-00008. PMID 10071668
- [Background] Ansink AC, Sie-Go DM, van der Velden J, Sijmons EA, de Barros Lopes A, Monaghan JM, Kenter GG, Murdoch JB, ten Kate FJ, Heintz AP. Identification of sentinel lymph nodes in vulvar carcinoma patients with the aid of a patent blue V injection: a multicenter study. Cancer. 1999 Aug 15;86(4):652-6. doi: 10.1002/(sici)1097-0142(19990815)86:43.0.co;2-r. PMID 10440693
- [Background] Rodier JF, Janser JC, Routiot T, David E, Ott G, Schneegans O, Ghnassia JP. Sentinel node biopsy in vulvar malignancies: a preliminary feasibility study. Oncol Rep. 1999 Nov-Dec;6(6):1249-52. doi: 10.3892/or.6.6.1249. PMID 10523690
- [Background] Kiss H, Ahner R, Hohlagschwandtner M, Leitich H, Husslein P. Fetal fibronectin as a predictor of term labor: a literature review. Acta Obstet Gynecol Scand. 2000 Jan;79(1):3-7. PMID 10646808
- [Background] Sideri M, De Cicco C, Maggioni A, Colombo N, Bocciolone L, Trifiro G, De Nuzzo M, Mangioni C, Paganelli G. Detection of sentinel nodes by lymphoscintigraphy and gamma probe guided surgery in vulvar neoplasia. Tumori. 2000 Jul-Aug;86(4):359-63. doi: 10.1177/030089160008600431. PMID 11016730
- [Background] Molpus KL, Kelley MC, Johnson JE, Martin WH, Jones HW 3rd. Sentinel lymph node detection and microstaging in vulvar carcinoma. J Reprod Med. 2001 Oct;46(10):863-9. PMID 11725728
- [Background] Sliutz G, Reinthaller A, Lantzsch T, Mende T, Sinzinger H, Kainz C, Koelbl H. Lymphatic mapping of sentinel nodes in early vulvar cancer. Gynecol Oncol. 2002 Mar;84(3):449-52. doi: 10.1006/gyno.2001.6572. PMID 11855886
- [Background] Hacker NF, Berek JS, Lagasse LD, Leuchter RS, Moore JG. Management of regional lymph nodes and their prognostic influence in vulvar cancer. Obstet Gynecol. 1983 Apr;61(4):408-12. PMID 6828268
- [Background] Moore RG, DePasquale SE, Steinhoff MM, Gajewski W, Steller M, Noto R, Falkenberry S. Sentinel node identification and the ability to detect metastatic tumor to inguinal lymph nodes in squamous cell cancer of the vulva. Gynecol Oncol. 2003 Jun;89(3):475-9. doi: 10.1016/s0090-8258(03)00130-6. PMID 12798714
- [Background] Moore RG, Granai CO, Gajewski W, Gordinier M, Steinhoff MM. Pathologic evaluation of inguinal sentinel lymph nodes in vulvar cancer patients: a comparison of immunohistochemical staining versus ultrastaging with hematoxylin and eosin staining. Gynecol Oncol. 2003 Nov;91(2):378-82. doi: 10.1016/j.ygyno.2003.07.006. PMID 14599869